CLINICAL TRIAL: NCT02666469
Title: Hyperbaric Oxygen and Focused Rehabilitation Program: A Feasibility Study in Improving Global Functioning After Stroke
Brief Title: HBOT Global Functioning After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Jo Carroll, Manager Anesthesia Research, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-8834-D
Record Dates: First submitted 2015-11-30; First posted 2016-01-28 (Estimated); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Stroke
Keywords: Hyperbaric oxygen treatment, rehabilitation
MeSH Terms: conditions — Stroke | interventions — Hyperbaric Oxygenation; Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A Hyperbaric Oxygen Therapy and Exercise Program (Active Comparator): Group A: Hyperbaric Oxygen Therapy (HBOT) and Exercise with HBOT sessions for 90 minutes, once daily, 5 times a week for 8 consecutive weeks. HBOT will be provided with 100% oxygen at 2.0 ATA. Patients will exercise in the multiplace hyperbaric chamber while receiving hyperbaric oxygen.
  Interventions: Other: Hyperbaric Oxygen Therapy (HBOT) and Exercise Program; Other: Exercise Program; Device: Hyperbaric Multiplace Chamber
- Group B Exercise Program (Active Comparator): Group B: Exercise Program in the hyperbaric medical unit without exposure to HBOT
  Interventions: Other: Exercise Program

INTERVENTIONS:
Other: Hyperbaric Oxygen Therapy (HBOT) and Exercise Program — HBOT provided with 100% oxygen at 2.0 ATA and rehabilitation program consisting of GRASP (60 min) and mental imagery (30 min)
  Arms: Group A Hyperbaric Oxygen Therapy and Exercise Program
Other: Exercise Program — Rehabilitation program consisting of GRASP (60 min) and mental imagery (30 min)
Device: Hyperbaric Multiplace Chamber — Patients will receive treatment in a multiplace Hyperbaric Chamber
  Arms: Group A Hyperbaric Oxygen Therapy and Exercise Program

SUMMARY:
Stroke is one of the leading causes of disability and death in North America and Europe. Up to 30% of stroke survivors never recuperate completely and suffer from loss of function and poor quality of life. To improve recovery after stroke, innovative interventions should be a priority.

Hyperbaric oxygen therapy (HBOT) is an intermittent inhalation of 100% oxygen in a hyperbaric chamber at a pressure higher than 1 absolute atmosphere (ATA). There is a growing body of evidence that HBOT can enhance ability of brain to changes its structure (neuroplasticity) in order to recover. Exercise program during HBOT can augment the effect. Although, recent randomized controlled trials in patients with chronic brain injury showed promising results, there are no studies demonstrating combine effect HBOT and exercise rehabilitation program on stroke recovery.

The proposed study investigates feasibility, safety and efficacy of using a combination of HBOT and exercise program to improve arm function recovery in chronic stroke patients. In this pilot randomized control trial, investigators will compare the combination of HBOT and the focused rehabilitation exercise program versus exercise program alone on recovery of arm function in patients with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* history of ischemic or hemorrhagic stroke 6-48 months confirmed by CT
* arm hemiparesis/hemiplegia
* Chedoke-McMaster Stroke Assessment Scale 3-6
* ability to follow verbal commands

Exclusion Criteria:

* women with positive pregnancy test or plans to become pregnant during the study period
* severe cognitive dysfunction (The Mini Mental State Examination <24 )
* claustrophobia
* seizure disorder
* active asthma
* severe chronic obstructive pulmonary disease
* history of spontaneous pneumothorax
* history of severe congestive heart failure with left ventricular ejection fraction < 30%; unstable angina
* myocardial infarction (within the last 3 months)
* chronic sinusitis
* chronic acute otitis media or major ear drum trauma
* current treatment with bleomycin, cisplatin, doxorubicin and disulfiram
* participation in another investigative drug or device trial currently or within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number or participants finishing the trial | 8 weeks
  The number of patients finishing the trial

SECONDARY OUTCOMES:
Total time spent doing rehabilitation exercise | 8 weeks
  Total time spent engaging in rehabilitation exercise (GRASP) in the trial

CONTACTS AND LOCATIONS:
Overall Officials: Rita Katznelson, MD, Principal Investigator — University Health Network, Toronto; Denyse Richardson, MD, Principal Investigator — Toronto Rehabilitation Institute, UHN
Locations (1):
- Toronto General Hospital, University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Schiavo S, Richardson D, Santa Mina D, Buryk-Iggers S, Uehling J, Carroll J, Clarke H, Djaiani C, Gershinsky M, Katznelson R. Hyperbaric oxygen and focused rehabilitation program: a feasibility study in improving upper limb motor function after stroke. Appl Physiol Nutr Metab. 2020 Dec;45(12):1345-1352. doi: 10.1139/apnm-2020-0124. Epub 2020 Jun 23. PMID 32574506